CLINICAL TRIAL: NCT04529811
Title: A Randomised, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Novel Rifaximin Formulations in Healthy Volunteers
Brief Title: Randomised, Placebo-controlled Safety and Pharmacokinetics Study of Novel Rifaximin Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBPK1001
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- Formulation 1 - Low Dose (Experimental): Rifaximin Formulation 1 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 1 Capsules - Mid Dose (Experimental): Rifaximin Formulation 1 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 1 Capsules - High Dose (Experimental): Rifaximin Formulation 1 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 1 Capsules - Max Dose (Experimental): Rifaximin Formulation 1 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 1 Capsules - Placebo (Placebo Comparator): Placebo Formulation 1 Capsules
  Interventions: Drug: Placebo
- Formulation 2 - Low Dose (Experimental): Rifaximin Formulation 2 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 2- Mid Dose (Experimental): Rifaximin Formulation 2 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 2 - High Dose (Experimental): Rifaximin Formulation 2 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 2 - Max Dose (Experimental): Rifaximin Formulation 2 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 2 - Placebo (Placebo Comparator): Placebo Formulation 2 Capsules
  Interventions: Drug: Placebo
- Formulation 3 - Low dose (Experimental): Rifaximin Formulation 3 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 3 - Mid dose (Experimental): Rifaximin Formulation 3 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 3 - High dose (Experimental): Rifaximin Formulation 3 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 3 - Max dose (Experimental): Rifaximin Formulation 3 Capsules
  Interventions: Drug: Rifaximin Novel Formulation
- Formulation 3 - Placebo (Placebo Comparator): Placebo Formulation 3 Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin Novel Formulation — Rifaximin Novel Formulation
  Arms: Formulation 1 - Low Dose; Formulation 1 Capsules - High Dose; Formulation 1 Capsules - Max Dose; Formulation 1 Capsules - Mid Dose; Formulation 2 - High Dose; Formulation 2 - Low Dose; Formulation 2 - Max Dose; Formulation 2- Mid Dose; Formulation 3 - High dose; Formulation 3 - Low dose; Formulation 3 - Max dose; Formulation 3 - Mid dose
Drug: Placebo — Placebo
  Arms: Formulation 1 Capsules - Placebo; Formulation 2 - Placebo; Formulation 3 - Placebo

SUMMARY:
Phase 1, Randomised, Placebo-Controlled, Single-Ascending Dose and Multiple-Dose with 3 novel RIFAXIMIN Formulations.

2 phases: Single-Ascending Dose (SAD) Phase and a Multiple-Dose (MD) Phase, Plus optional open-label, crossover Food Effect (FE) Evaluation

Primary objective: evaluate the safety and tolerability of three novel formulations of rifaximin in healthy volunteers.

Secondary objective: evaluate the pharmacokinetics (PK) of the novel formulations and to assess for the presence of exploratory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* The participant has the ability and willingness to sign a written informed consent, is either male or female aged between 18 and 65 years, inclusive, at the time of informed consent, is in good general health, and has a body mass index (BMI) at least 18 kg/m2 and at most 34 kg/m2, and a minimum body weight of 45 kg.
* The participant must have suitable venous access for blood sampling and be able and willing to complete the study and comply with all study instructions and attend the necessary visits.
* A negative pregnancy test is required for all women of child-bearing potential (WOCBP). WOCBP and men must agree to use highly effective contraception methods from screening through the end of the study. Follicle stimulating hormone (FSH) testing will be conducted for post-menopausal women without surgical evidence of sterility (total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).

Exclusion Criteria:

* Female participant who is pregnant, trying to become pregnant, or breast feeding.
* Participant with a known or suspected intolerance to rifaximin or the excipients used in the novel formulations.
* Participant has had any major illness or systemic infection (including COVID [coronavirus disease] -19) within 4 weeks of the Screening Visit or has a clinically relevant history or currently suffering from any disease or condition that, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk. Participant has liver function tests >1.1x the upper limit of normal or any other abnormal laboratory test that the Investigator deems as clinically significant.
* Participant has human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection, a clinically relevant history of or current evidence of abuse of alcohol or other drugs. Participant is currently a tobacco smoker or was a tobacco smoker within 6 months of the Baseline Visit.
* Participant has received any investigational product within 4 weeks or 5 half-lives of the product, whichever is greater, prior to the Baseline Visit or is scheduled to receive an investigational product (other than the study product) or is scheduled for a medical procedure during the study period. Participant is taking probiotics.
* Participant is taking any medications which are known cytochrome P450 3A (CYP3A) or P-glycoprotein (Pgp) inhibitors/inducers or is currently using any medication that, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events | Up to 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schwabe, MD, Principal Investigator — Auckland Clinical Studies
Locations (1):
- Auckland Clinical Studies, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No